CLINICAL TRIAL: NCT01615250
Title: Phase I Study to Evaluate the Efficacy and Safety of Intramyocardial Implantation of Peripheral Mononuclear Cells With CD34+ Stem Cells in Patient With Ischemic Cardiomyopathy After Preparatory Course of Shock - Wave Therapy
Brief Title: Implantation of Peripheral Stem Cells in Patient With Ischemic Cardiomyopathy
Acronym: ISCIC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odessa National Medical University (Other)
Responsible Party: Principal Investigator, Iurii Kozlov, Dr., PhD Iurii I Karpenko, Odessa National Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCIC-2012
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Standard therapy (No Intervention): Treatment with standard therapy. Cardiospec shock-wave therapy
- Stem cells (Active Comparator): Group of of intramyocardial implantation of peripheral mononuclear cells with CD34+ stem cells in patient with ischemic cardiomyopathy after preparatory course of shock - wave therapy.
  Interventions: Biological: Intramyocardial implantation of stem cells

INTERVENTIONS:
Biological: Intramyocardial implantation of stem cells — Intramyocardial implantation of autologous peripheral mononuclear cells with CD34+ stem cells by NOGA.XP navigation system. Сell concentration is 200 million cells in 1 ml.
  Arms: Stem cells

SUMMARY:
This is a randomized study of efficiency and safety of intramyocardial implantation of peripheral mononuclear cells with high concentration of CD34+ stem cells in patients with myocardial ischemia after preparatory course of shock - wave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic cardiomyopaty and HF II-IV NYHA class
* MI more than 6 months before the study
* LVEF less than 35%
* Absence effect of coronary revascularization during 6 months
* Optimal pharmacological therapy no less than 8 weeks
* Heart transplantation is contraindicated
* Patients with implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D)
* Patients giving informed consent

Exclusion Criteria:

* Acute coronary syndrome
* Coronary revascularization less than 6 months
* Patients requiring surgical correction of post-MI aneurism
* LV wall thickness less than 5 mm in site of possible injection
* Patients with CRT implanted within 3 month before cells injection
* Clinically significant associated diseases
* Active oncology desiase
* Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction and regional wall motion score index | 6 and12 months
  Change in global left ventricular ejection fraction and regional wall motion score index.

SECONDARY OUTCOMES:
Incidence of the major adverse cardiac events | 6 and 12 months
  Incidence of the major adverse cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Iurii I Karpenko, Dr, PhD, Principal Investigator — Odessa National Medical University
Locations (1):
- Odessa Regional Clinical Hospital, Odesa, Ukraine